CLINICAL TRIAL: NCT04309643
Title: A Phase 1, Open-label Study to Assess the Effect of CTP-543 on the Pharmacokinetics of Oral Contraceptives in Healthy Adult Female Subjects
Brief Title: Drug-drug Interaction Study of CTP-543 and Oral Contraceptives in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CP543.1005
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Healthy Volunteers
Keywords: Oral contraceptive; Drug-drug Interaction; CTP-543
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTP-543 (Experimental): In Period 1, participants will receive a single oral dose of the combination oral contraceptive (OC) on Day 1. There will be a washout period of 7 days between dosing in Period 1 and the first dose in Period 2. In Period 2, participants will receive twice daily oral doses of CTP-543 for 8 consecutive days with a single dose of the combination OC co-administered on Day 4.
  Interventions: Drug: CTP-543; Drug: Combined oral contraceptive containing Ethinyl estradiol (EE) and Levonorgestrel (LNG)

INTERVENTIONS:
Drug: CTP-543 — Investigational Drug
Drug: Combined oral contraceptive containing Ethinyl estradiol (EE) and Levonorgestrel (LNG) — Oral contraceptive in the form of 1 fixed combination tablet of Seasonique or generic equivalent (0.03 mg EE / 0.15 mg LNG)

SUMMARY:
This is a Phase 1, fixed sequence, multiple dose, open-label study of the effect of CTP-543 on oral contraceptive pharmacokinetics in healthy female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female participants of non-childbearing potential, or adult females of childbearing potential who agree to use birth control methods described in the protocol
* If of reproductive age, willing and able to use a medically highly effective form of birth control 28 days prior to first dose, during the study and for 28 days following last dose of study medication. Examples of medically highly effective forms of birth control are:

  1. Surgical sterilization of the partner (via vasectomy, hysterectomy, bilateral tubal ligation or bilateral salpingectomy) at least 4 months prior to first dose or post-menopausal with amenorrhea for at least 1 year prior to the first dosing and follicle-stimulating hormone (FSH) serum levels (> 40 IU/L) consistent with postmenopausal status
  2. Sexual partner is sterile, or of the same sex
  3. Double-barrier method (any combination of physical and chemical methods)
  4. Non-hormone releasing intrauterine device in females
* Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dosing and throughout the study
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2
* Medically healthy with no clinically significant medical history, physical examination, laboratory tests, vital signs, or ECGs
* Understands the study procedures in the informed consent form, and be willing and able to comply with the protocol

Exclusion Criteria:

* Positive pregnancy test
* History or presence of clinically significant medical or psychiatric condition or disease
* History of any illness that might confound the results of the study or pose an additional risk to the subject by their participation in the study
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing
* A positive tuberculosis test at screening or history of incompletely treated or untreated tuberculosis
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Donation of blood or significant blood loss within 56 days prior to dosing

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
AUC0-t | From the start of Period 1 to completion of Period 2 (16 days)
  Area Under the Plasma Concentration-Time Profile
AUC0-inf | From the start of Period 1 to completion of Period 2 (16 days)
  Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time
Cmax | From the start of Period 1 to completion of Period 2 (16 days)
  Maximum observed concentration of drug in plasma

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 58 days
  An adverse event is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention
Number of Participants With Clinically Significant Change in Vital Signs | Up to 44 days
  Blood pressure, heart rate, respiratory rate, and temperature
Number of Participants With Clinically Significant Change in Clinical Laboratory Evaluations | Up to 44 days
  Hematology, serum chemistry, coagulation, and urinalysis
Number of Participants With Clinically Significant Change to the Physical Examination | Screening (Day -28)
  Symptom-driven physical examinations may be performed at other times, if deemed necessary
Number of Participants With Clinically Significant Change in Electrocardiogram | Up to 40 days
  12-Lead ECG

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Inc., Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No